CLINICAL TRIAL: NCT06365528
Title: Tunneled Versus Non-Tunneled Peripherally Inserted Central Catheter and Their Effects on Reducing Combined or Isolated Outcomes (Obstruction, Infection, Thrombosis, and Dislodgement): Multicenter Randomized Clinical Trial
Brief Title: Tunneled Peripherally Inserted Central Catheter (PICC) in Adult Patients and Associated Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Hospital Moinhos de Vento (Other); Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023-0232
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: CLABSI - Central Line Associated Bloodstream Infection; Deep Vein Thrombosis; Dislodged Catheter; Occlusion; Catheter Rupture; Catheter (Other); Complications
MeSH Terms: conditions — Venous Thrombosis; Bites and Stings

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Prospective Randomized Open, Blinded End-point (PROBE Study)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tunneled PICC (Experimental): The intervention group will consist of adult patients who will have PICCs inserted using the catheter tunneling technique. The technique involves the catheter being exteriorized through the skin at a site different from the blood vessel puncture site, thus traversing a subcutaneous tunnel.
  Interventions: Procedure: Subcutaneous tunnelling
- Non-tunneled PICC (Active Comparator): The control group will consist of adults patients who will have PICCs inserted using the conventional technique
  Interventions: Procedure: Non-tunnelling

INTERVENTIONS:
Procedure: Subcutaneous tunnelling — The Subcutaneous tunnelling group will undergo PICC placement under ultrasonography. Procedures will be implemented under hand hygiene, maximal sterile barrier, and chlorhexidine. The targeted arm will be sterilized with a mixture of chlorhexidine and isopropyl alcohol, and a sterile drape will be placed to cover the entire procedure feld from head to toe and place with additional subcutaneous tunnelling. After vein puncture with the access needle, a Nitinol guidewire will be placed as usual. We will make a tunnel distal to the initial venepuncture site using an additional 14-gauge needle. After resolution of the loop over the venepuncture site, a peel-away sheath will be placed over the wire. The catheter will be trimmed to the distance between the venepuncture site and cavoatrial junction plus the subcutaneous tunnel before being inserted in the usual manner.
  Arms: Tunneled PICC
Procedure: Non-tunnelling — The Non-tunnelling group will have PICC placement with the traditional method under ultrasonography. Procedures will be implemented under hand hygiene, maximal sterile barrier, and chlorhexidine. The targeted arm will be sterilized with a mixture of chlorhexidine and isopropyl alcohol, and a sterile drape will be placed to cover the entire procedure feld from head to toe. After vein puncture with the access needle, a Nitinol guidewire will be placed. After, a peel-away sheath will be placed over the wire. The catheter will be trimmed to the distance between the venepuncture site and cavoatrial junction.
  Arms: Non-tunneled PICC

SUMMARY:
The aim of this multicenter randomized clinical trial is to compare the tunneling technique of PICC insertion with the non-tunneled insertion technique in the incidence of the combined or isolated outcome of catheter-related bloodstream primary infection, thrombosis, obstruction, and accidental dislodgement in the adult population within a period of up to 30 days.

DETAILED DESCRIPTION:
The data published this year from a multicenter study in Brazil presenting the patterns of use and clinical outcomes of PICC indicated that centers with vascular access teams, adoption of best practices, and current technologies result in low rates of complications, such as primary bloodstream infections related to the catheter, deep vein thrombosis, and reversible occlusion. Despite these more recent data showing that complications related to PICC can be mitigated by the use of technology, vascular access teams, adoption of best practices, and infection control measures, there is still room to incorporate new techniques in PICC insertion with the aim of further reducing avoidable complications. For example, recent studies with robust methodology have demonstrated the benefit of the tunneling technique compared to the conventional insertion technique. A randomized clinical trial showed that the dwell time of the device inserted using the tunneling technique was longer compared to the conventional technique without tunneling in adult patients, along with a lower incidence of thrombosis and infection. At the Hospital de Clínicas de Porto Alegre, recently, nurses from the PICC Team were trained in the tunneling technique at a reference center in Brazil. The initial results of tunneling in adult, pediatric, and neonatal patients are encouraging.

The observed results of implementing the technique indicate that there is potential to reduce avoidable complications and prompt us to propose a multicenter randomized controlled trial involving two additional institutions with similar profiles regarding the composition of Vascular Access Teams, adoption of best practices related to catheter care, and active ongoing education. To our knowledge, robust studies of this nature are not currently being conducted in Brazil.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (>= 18 years old) admitted to medical clinics, surgical clinics, or ICU, who have an indication for PICC insertion;

Exclusion Criteria:

* patients with Chronic Kidney Disease, whether dialytic or not;
* patients in critical or unstable condition characterized by the need for intubation, respiratory rate <8 or >35 breaths per minute, oxygen saturation <90%, heart rate <40 or >140 beats per minute, systolic blood pressure <90mmHg, decreased Glasgow Coma Scale >2 points, or prolonged (>5 minutes) or repeated seizures;
* patients with cognitive deficits that impair their understanding of the study and do not have a responsible party to assist in this stage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
End of therapy or catheter removal free from complications | Up to 30 days
  Time in days

CONTACTS AND LOCATIONS:
Overall Officials: Eneida R Rabelo da Silva, ScD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Brazil

IPD SHARING:
Plan to Share IPD: No